CLINICAL TRIAL: NCT05125406
Title: Prevention of ICU-Related Anxiety in Lung Transplantation by Virtual Reality Therapy - PIRAT Study
Acronym: PIRAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-16
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Transplantation, Lung; Depression, Anxiety; PTSD
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic | interventions — Implosive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exposure therapy using Virtual Reality (ETVR) (Experimental)
  Interventions: Behavioral: Exposure therapy with Virtual Reality.
- No exposure therapy with Virtual Reality. (No Intervention)

INTERVENTIONS:
Behavioral: Exposure therapy with Virtual Reality. — Experimental arm patients will be offered Exposure therapy with Virtual Reality (ETRV) support with a virtual reality headset. A scenario with progressively increasing stress levels linked to the ICU environment and different situational contexts (alarms, etc.) will be presented to patients. This habituation to the potentially anxiety context of ICU will reduce the occurrence of psycho-cognitive disorders by progressive extinction phenomenon.
  Arms: Exposure therapy using Virtual Reality (ETVR)

SUMMARY:
ICU patients frequently face complicated recovery processes, including long-term anxiety disorders. Lung transplantation (LTx) offers people with terminal respiratory conditions both the hope of prolonged survival and a better quality of life related to health. Among the disorders usually encountered in the postoperative period of LTx are anxio-depressive disorders. These anxiety disorders affect the quality of life related to health and compromise the follow-up of the patient by phenomenon of psychological disinvestment. Other psychological disorders are also anchored in the patient's experience of this post-surgical ICU period (ie, depressive episodes and/or, at a distance, post-traumatic stress disorder (PTSD). Various models of management of anxio-depressive disorders and PTSD are proposed in the literature. To our knowledge, while many of them have shown their efficiency in the curative management of disorders, few have demonstrated their effectiveness in preventing them. Exposure therapies using virtual reality (ETVR) have in the past demonstrated their effectiveness in many areas of psychiatry. In our study, experimental arm patients will be offered ETRV support with a virtual reality headset. A scenario with progressively increasing stress levels linked to the ICU environment and different situational contexts (alarms, etc.) will be presented to patients. This habituation to the potentially anxiety context of ICU will reduce the occurrence of psycho-cognitive disorders by progressive extinction phenomenon.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Registration on the lung transplant waiting list
* Signature of consent

Exclusion Criteria:

* Minor patient, pregnant or breastfeeding woman, or not affiliated to the social security scheme
* Patient under guardianship or curatorship
* Patient with a history of mental illness
* Patient not mastering the French language
* Patient deprived of liberty
* Patient carrying a transplanted organ (liver, kidney, heart ...)
* Lung re-transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Spielberger state trait anxiety inventory for adults | Post-transplant
  The State-Trait Anxiety Inventory (STAI) has been used extensively in research and clinical practice. It comprises separate self-report scales for measuring state and trait anxiety. The S-Anxiety scale (STAI Form Y-1) consists of twenty statements that evaluate how respondents feel "right now, at this moment." The T-Anxiety scale (STAI Form Y-2) consists of twenty statements that assess how people generally feel.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression scale (HADS) | Post-transplant
  The Hospital Anxiety and Depression Scale (HADS) measure anxiety and depression in a general medical population of patients.
The Impact of Event Scale -Revised | Post-transplant
  The IES-R is a solid measure of post-trauma phenomena and Posttraumatic Stress Disorder.
Post-traumatic stress disorder Checklist Scale (PCLS) | Post-transplant
  The IES-R is a solid measure of post-trauma phenomena and Posttraumatic Stress Disorder.

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Des Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided